CLINICAL TRIAL: NCT01721395
Title: Effect of Agave Syrup, Placebo, and No Treatment on Nocturnal Cough and Sleep Quality for Coughing Infants/Toddlers and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Zarbee's Inc. (Industry)
Responsible Party: Principal Investigator, Ian M. Paul, M.D., M.Sc., Professor of Pediatrics and Public Health Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB001
Record Dates: First submitted 2012-10-26; First posted 2012-11-05 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Cough
Keywords: Cough; Nocturnal Cough; Agave; Sleep Quality; Childhood cough
MeSH Terms: conditions — Cough; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Colored, Flavored water (Placebo Comparator): The placebo will be colored to approximate the reddish amber color of the agave syrup. The placebo will use the same flavoring used in the agave syrup. The placebo will be created in a GMP facility
  Interventions: Dietary Supplement: Agave Syrup
- Agave Syrup (Experimental): The formulation of pasteurized agave syrup consists of pasteurized agave syrup and natural flavoring.
  Interventions: Dietary Supplement: Agave Syrup
- Air-filled oral syringe (Sham Comparator): Air-filled oral syringe to match experimental and placebo arm
  Interventions: Dietary Supplement: Agave Syrup

INTERVENTIONS:
Dietary Supplement: Agave Syrup
  Other Names: Zarbee's Naturals Agave Baby Cough Syrup

SUMMARY:
Cough is a frequent symptom in children and infants and is one of the most common reasons parents visit a healthcare provider for their child. The US Food and Drug Administration has issued a warning that over-the-counter cough and cold medicines including antihistamines, decongestants, anti-tussives, and expectorants should not be administered to children younger than 2 years of age due not only to lack of proven efficacy, but also because of important safety concerns. Honey, another method of soothing cough cannot be used in children <1 year due to concerns for infantile botulism. A preparation from agave syrup has been created to address the need for an infant cough syrup. Although no studies have formally evaluated the use of agave nectar for nocturnal cough associated with Upper Respiratory Infections, the demulcent effect and sweet taste of agave nectar may provide some relief from cough in children.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male or female infant who is 2 to <48 months of age.
* presents with a non-specific acute cough for 7 or fewer days' duration.
* Parents/legal authorized representative reporting at least moderate cough and cold symptoms.
* Parent/legal authorized representative was in the home with the child on the night prior to enrollment and plans to be in the home with the child on the night when study treatment will be administered
* Parent/legal authorized representative who is willing and able to comply with study requirements.

Exclusion Criteria:

* Previous participation in this clinical trial
* Gestational age at birth <35 weeks.
* Signs or symptoms of a more treatable disease (eg, asthma, pneumonia, laryngotracheobronchitis, sinusitis, allergic rhinitis).
* Diagnosis of influenza, bronchiolitis or respiratory syncytial virus (RSV).
* History of reactive airways disease, asthma, or chronic lung disease.
* Use of any medication or honey to treat cough within 6 hours of bedtime on the evening prior to or on the day of enrollment.
* Presence of any significant disease including immunodeficiency, hepatic, renal,cardiovascular, or hematologic disease or any other health condition that, in the opinion of the investigator, would preclude participation in the study.
* Known allergy to agave nectar or grape flavoring

Ages: 2 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Efficacy:Change in Cough Frequency based on parent responses to the Pediatric Cough Questionnaire | Baseline (night 1) and End of night 2
  Change from baseline in cough frequency between the first night and the end of the second night. Parents/caregivers will complete a Pediatric Cough Questionnaire (a subjective parent report of cough) using a 0-6 point Likert scale with 0=not at all to 6=extremely often to assess frequency of cough. The same parent/caregiver that completed the questionnaire in the clinic will be asked to complete the questionnaire during the follow-up telephone call.

SECONDARY OUTCOMES:
Efficacy: Change in Response to Other symptom responses on the Pediatric Cough Questionnaire(parental report) | Change from Baseline (night 1) to End of Second Night
  Change from baseline (night 1) and the end of the second night for each of the remaining questionnaire items pertaining to cough and cold symptoms and the symptoms affect on sleep.
  Parents/caregivers will complete a Pediatric Cough Questionnaire (a subjective parent report of cold symptoms) using a 0-6 point Likert scale with 0=not at all to 6=extremely often to assess cold symptoms.
  * severity of cough
  * bothersome nature of cough
  * how much the cough affected the child's and parent's/caregiver's ability to sleep
  * severity of stuffy nose
  * severity of runny nose The same parent/caregiver that completed the questionnaire in the clinic will be asked to complete the questionnaire during the follow-up telephone call.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State University
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Beiler JS, Vallati JR, Duda LM, King TS. Placebo effect in the treatment of acute cough in infants and toddlers: a randomized clinical trial. JAMA Pediatr. 2014 Dec;168(12):1107-13. doi: 10.1001/jamapediatrics.2014.1609. PMID 25347696